CLINICAL TRIAL: NCT01142687
Title: Effects of Dihydrocapsiate on Adaptive and Diet-Induced Thermogenesis Following 4 Weeks of Very Low Calorie Diet
Brief Title: Effects of Dihydrocapsiate on Adaptive and Diet-Induced Thermogenesis With a High Protein Very Low Calorie Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 08-05-113
Record Dates: First submitted 2010-06-10; First posted 2010-06-11 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Healthy
Keywords: Resting energy expenditure (REE); metabolic rate
MeSH Terms: interventions — capsiate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- dihydrocapsiate 3 mg (Active Comparator): • Group 1: 1 Dihydrocapsiate capsule and 2 placebo capsules three times a day within 30 minutes before breakfast, lunch and dinner
  Interventions: Dietary Supplement: dihydrocapsiate capsule
- dihydrocapsiate 9 mg (Active Comparator): • Group 2: 3 Dihydrocapsiate capsules three times per day within 30 minutes before breakfast, lunch and dinner
  Interventions: Dietary Supplement: dihydrocapsiate capsule
- Placebo capsule (Placebo Comparator): • Group 3: 3 placebo capsules three times per day within 30 minutes before breakfast, lunch and dinner
  Interventions: Dietary Supplement: dihydrocapsiate capsule

INTERVENTIONS:
Dietary Supplement: dihydrocapsiate capsule — * Group 1: 1 dihydrocapsiate capsule and 2 placebo capsules three times a day within 30 minutes before breakfast, lunch and dinner.
  * Group 2: 3 dihydrocapsiate capsules three times per day within 30 minutes before breakfast, lunch and dinner
  * Group 3: Placebo 3 capsules three times per day within 30 minutes before breakfast, lunch and dinner
  Other Names: chili pepper

SUMMARY:
The study is designed to determine the effects of a non-pungent supplement from sweet chilli pepper on resting metabolic rate and diet-induced thermogenesis (DIT) after a period of very low calorie intake over 4 weeks.

DETAILED DESCRIPTION:
Thirty-six subjects will be recruited by public advertisement. Postmenopausal women and men over age 30 with a body mass index (BMI) between 27 to 35 kg/m2,and in good health by history, physical examination, and basic laboratory screening (complete blood count, serum chemistries, liver panel, and lipid panel) will be selected for study. Subjects with type 2 diabetes or glucose intolerance will be excluded as will individuals who regularly drink more than one alcoholic beverage daily. Thirty-six men and women who meet the selection criteria below will be randomly assigned to one of three arms providing CH-19 at two dose levels per day vs. placebo capsules.

This will be a prospectively randomized double blind study in which neither the subjects nor the clinical research personnel will be aware of whether the subjects will be assigned to placebo or dihydrocapsiate at two different doses. A total of 36 subjects will be divided among three groups.

To keep the number of capsules taken by each subject constant, all subjects will take three capsules three times per day containing the appropriate number of active or placebo capsules and will be randomized after screening to one of three groups:

* Group 1: Dihydrocapsiate 1 capsule and 2 placebo capsules three times a day within 30 minutes before breakfast, lunch and dinner.
* Group 2: Dihydrocapsiate 3 capsules three times per day within 30 minutes before breakfast, lunch and dinner
* Group 3: Placebo 3 capsules three times per day within 30 minutes before breakfast, lunch and dinner

ELIGIBILITY:
Inclusion Criteria:a.

1. Postmenopausal female or male over 30 years of age at the time the consent form is signed.
2. Subject has a BMI between 27 and 35 kg/m2
3. Subject is in good health based on history, physical examination, and basic laboratory studies.
4. Consumes less than one alcoholic beverage per day
5. Is a non-smoker for at least three months
6. Willing to follow a Very Low Calorie Diet of 800 calories per day using meal replacements
7. Ethical: Subject must sign the Institutional Review Board-approved written informed consent prior to the initiation of any study specific procedures or randomization. A subject will be excluded for any condition that might compromise the ability to give truly informed consent for participation in the study.

Exclusion Criteria:

1. Any subject with known allergy to chili peppers by history.
2. Any subject with type 2 diabetes or glucose intolerance
3. Consumes more than one alcoholic beverage per day
4. Any subject participating in regular vigorous exercises other than ordinary daily walks or who is unwilling to maintain their usual level of exercise during the study.
5. Any subject with a diagnosed eating disorder or who is addicted to any medications.
6. Any subject currently taking antidepressants or weight loss medication.
7. Any subjects with a history of gastrointestinal surgery, uncontrolled hypertension, or other serious medical condition, such as chronic hepatitis or renal disease, bleeding disorder, congestive heart disease, chronic diarrhea disorders, myocardial infarction, coronary artery bypass graft, angioplasty within 6 months prior to screening, current diagnosis of uncontrolled hypertension (defined as BP >160mmHg, diastolic BP>95mmHg), active or chronic gastrointestinal disorders, bulimia, anorexia, laxative abuse, or endocrine diseases (except thyroid disease requiring medication) as indicated by medical history or routine physical examination.
8. Major surgery within 12 weeks prior to subject randomization and/or screening, especially cardiac surgery
9. Is currently a smoker who has a therapeutic plan to quit smoking anytime during the study period; or if not a current smoker, has quit smoking within the past 3 months.
10. Known HIV positive.
11. Clinical evidence of current malignancy with the exception of basal cell or squamous cell carcinoma of the skin and cervical intraepithelial neoplasia.
12. Currently receiving systemic chemotherapy and/or radiotherapy.
13. Active bleeding.
14. Subject has any disorder including illiteracy or visual impairment that compromises the ability of the subject to give written informed consent and/or to comply with study procedures.
15. In the opinion of the study investigator has a risk of non-compliance with study procedures, or cannot read, understand or complete study related materials.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2008-11; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Adaptive Thermogenesis | 4 weeks
  To determine the effects of dihydrocapsiate at two doses on the decrease in resting metabolic rate which occurs after a period of very low calorie intake over 4 weeks

SECONDARY OUTCOMES:
Diet-Induced thermogenesis | 4 weeks
  To determine the effects of dihydrocapsiate at two doses on diet-induced thermogenesis (DIT) following a 426 Calorie high protein liquid meal

CONTACTS AND LOCATIONS:
Overall Officials: David Heber, MD, PhD, Principal Investigator — University of California, Los Angeles

REFERENCES:
- [Result] Lee TA, Li Z, Zerlin A, Heber D. Effects of dihydrocapsiate on adaptive and diet-induced thermogenesis with a high protein very low calorie diet: a randomized control trial. Nutr Metab (Lond). 2010 Oct 6;7:78. doi: 10.1186/1743-7075-7-78. PMID 20925950